CLINICAL TRIAL: NCT04029818
Title: Preliminary Study to Evaluate the Effect of the Consumption of Bifidobacterium BSL_PS404 on LDL-cholesterol Levels in Healthy Volunteers
Brief Title: Evaluation of a Probiotic on LDL-cholesterol Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P046
Record Dates: First submitted 2019-07-22; First posted 2019-07-23 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-07

CONDITIONS: Cardiovascular Diseases; LDL-cholesterol
Keywords: LDL-cholesterol; Probiotics
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Volunteers will take a capsule with Bifidobacterium BSL_PS404 (3x109 cfu) daily.
  Interventions: Biological: Bifidobacterium BSL_PS404
- Placebo (Placebo Comparator): Volunteers will take a capsule with maltodextrin daily.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Bifidobacterium BSL_PS404 — Each participant will consume 1 capsule daily at lunch for 8 weeks.
  Arms: Probiotic
Biological: Placebo — Each participant will consume 1 capsule daily at lunch for 8 weeks.
  Arms: Placebo

SUMMARY:
The aim of the present study is to evaluate the ability of Bifidobacterium BSL_PS404 in reducing LDL-cholesterol levels in healthy individuals.

DETAILED DESCRIPTION:
There is a strong correlation between LDL-cholesterol and cardiovascular diseases.

Conjugated bile acids help to break down and emulsify dietary fat into micelles that promote their absorption by the enterocytes. The disruption or alteration of these micelles may interfere with the absorption of cholesterol.

Several intestinal bacteria strains are capable of carrying out numerous biotransformations of bile salts during their enterohepatic circulation, such as the hydrolysis of the conjugated bile acids by the action of hydrolases. The mechanism proposed to explain the cholesterol-lowering activity of these probiotic strains is that, due to the greater bile salt hydroxylation in the intestine, the formation of micelles would decrease and, therefore, the absorption of cholesterol and lipids would be decrease too. In addition, probiotics may also increase the excretion of bile acids in the stool, possibly by binding or absorbing them. This increase in fecal secretion of bile acids would require an increase in the hepatic catabolism of cholesterol for the synthesis of bile acids. All these processes may help to reduce LDL-cholesterol levels Bifidobacterium BSL_PS404 is a bacterium isolated from maternal milk with QPS category that presents a high hydrolase activity that exceeds in more than 20% the activity of other reference strains.

ELIGIBILITY:
Inclusion Criteria:

* Levels of LDL-cholesterol between 100 and 190 mg/dL.
* Accept freely to participate in the study and sign the informed consent document.

Exclusion Criteria:

* Be pregnant.
* Have planned to carry out a dietary intervention or exercise practice with the aim of losing weight in the coming weeks.
* Having a serious illness.
* Having diabetes.
* Having a cerebrovascular disease.
* Being allergic to any group of antibiotics.
* Take probiotics in the form of supplements at least 4 weeks before.
* Take antibiotics at least 4 weeks before.
* Being taking products or drugs to control cholesterol levels

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol | 8 weeks
  Levels of LDL-cholesterol in plasma

SECONDARY OUTCOMES:
Total cholesterol | 8 weeks
  Levels of total cholesterol in plasma
HDL-cholesterol | 8 weeks
  Levels of HDL-cholesterol in plasma
Triglycerides | 8 weeks
  Levels of triglycerides in plasma
Glucose | 8 weeks
  Levels of glucose in plasma
Blood pressure | 8 weeks
  Systolic and diastolic pressure
Body mass index | 8 weeks
  A person's weight in kilograms (kg) divided by his or her height in meters squared

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Quesada, MD, PhD, Study Chair — Medical specialist in Endocrinology, Hospital San Cecilio de Granada
Locations (1):
- Hospital San Cecilio, Granada, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No